CLINICAL TRIAL: NCT05600556
Title: The Role of Virtual Reality (VR) in Patient Experience When Used for Magnetic Resonance-Guided Radiation Therapy (MRgRT)
Brief Title: Virtual Reality for the Improvement of Patients Understanding of Disease and Treatment (MRgRT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: ViewRay (funding sponsor) bankruptcy
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 22C.714; JT 20764 (Other: JeffTrial Number)
Record Dates: First submitted 2022-10-18; First posted 2022-10-31 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Magnetic Resonance Spectroscopy; X-Rays; Practice Guidelines as Topic; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort I (standard imaging) (Active Comparator): Patients receive 2D image review using standard computer screen on study. Patients undergo MRI and CT imaging at screening and on study
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Other: Best Practice; Other: Questionnaire Administration
- Cohort II (virtual reality) (Experimental): Patients receive image review using virtual reality stimulation on study. Patients also view MRI treatment room using virtual reality stimulation. Patients undergo MRI and CT imaging at screening and on study
  Interventions: Procedure: Magnetic Resonance Imaging; Procedure: Computed Tomography; Other: Virtual Technology Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
  Arms: Cohort I (standard imaging)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
  Arms: Cohort I (standard imaging)
Other: Best Practice — Review imaging on standard computer screen
  Other Names: standard of care; standard therapy
  Arms: Cohort I (standard imaging)
Other: Questionnaire Administration — Complete questionnaire
  Arms: Cohort I (standard imaging)
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging Scan; Medical Imaging; Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; NMR Imaging; NMRI; nuclear magnetic resonance imaging
  Arms: Cohort II (virtual reality)
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; computerized axial tomography; Computerized Tomography; CT; CT SCAN; tomography
  Arms: Cohort II (virtual reality)
Other: Virtual Technology Intervention — Review virtual reality images
  Other Names: Virtual Reality Intervention; Virtual Technology
  Arms: Cohort II (virtual reality)
Other: Questionnaire Administration — Complete questionnaire
  Arms: Cohort II (virtual reality)

SUMMARY:
This clinical trial explores if using virtual reality (VR) headsets will help to improve patient understanding of their disease and decrease anxiety about treatment. Three-dimensional (3D) images may help the patient visualize their tumor and location better and therefore understand potential side effects. Visualizing a virtual representation of the magnetic resonance imaging (MRI) linear accelerator (Linac) may decrease treatment related anxiety.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Examine patient reported comprehension of their tumor characteristics and treatment plan following 3D virtual reality review of their imaging.

SECONDARY OBJECTIVE:

I. Examine patient reported treatment related anxiety prior to and following virtual reality (VR) simulation of the MRI Linac treatment process.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive two-dimensional (2D) image review using standard computer screen on study. Patients undergo MRI and computed tomography (CT) imaging at screening and on study.

COHORT II: Patients receive image review using virtual reality stimulation on study. Patients also view MRI treatment room using virtual reality stimulation. Patients undergo MRI and CT imaging at screening and on study.

ELIGIBILITY:
Inclusion Criteria:

* Age: above 18 years
* Participants must be histologically proven neoplasm
* Planned to undergo radiation treatment using the MR Linac

Exclusion Criteria:

* Inability to tolerate virtual reality headset
* Non-English speaking patients
* Pediatric patients are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Increase in composite knowledge questionnaire score | At Baseline
  Pre- and post-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.
Increase in composite knowledge questionnaire score | At first on treatment visit (after starting radiation)
  Pre- and post-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.

SECONDARY OUTCOMES:
General anxiety | At Baseline
  Pre-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.
General anxiety | At first on treatment visit (after starting radiation)
  Post-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.
MRI specific anxiety | Baseline and after MRI scan at time of planning scan
  Pre- and post-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.
Plan review understanding | Baseline and at first on treatment visit (after starting radiation)
  Pre- and post-intervention knowledge summary scores and anxiety scores will be summarized using means, standard deviations, and ranges. Average change will be estimated for each group along with 95% confidence intervals and the difference between groups will be estimated with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Mueller, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States